CLINICAL TRIAL: NCT02156934
Title: Evaluation the Effect of Autologous Muscle Derived Stem Cells Injection Into the Paraurethral Tissues for Treatment of Stress Urinary Incontinency,The Randomized Clinical Trial Phase II
Brief Title: Paraurethral Transplantation of Autologous Muscle Derived Stem Cells for Treatment of Stress Incontinency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Kidney-002
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Stress Urine Incontinency
Keywords: autologous stress urinary incontinence muscle derived cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muscle derived stem cell (Experimental): Paraurethral injection of muscle derived stem cell in patients with stress urine incontinency.
  Interventions: Biological: paraurethral injection

INTERVENTIONS:
Biological: paraurethral injection — Paraurethral injection of muscle derived stem cell in patients with stress urine incontinency.

SUMMARY:
This study was designed to provide confirmation of efficacy of muscle derived stem cells (MDCs) for the treatment of SUI in women.

DETAILED DESCRIPTION:
The investigators will be assessed the 12-month potential efficacy of autologous muscle derived cells as therapy for stress urinary incontinence. A total of 20 women in whom stress urinary incontinence had not improved underwent intra-sphincter injection of low doses 50×106 of autologous muscle derived cells, which will be derived from biopsies of their deltoid muscle. Assessments will be made at 1, 3, 6 and 12 months after cell injection. Changes in stress urinary incontinence severity were evaluated by pad test, diary of incontinence episodes and quality of life surveys.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Stress Urinary Incontinence symptoms
* Urodynamic stress incontinence confirmed with multichannel urodynamic testing
* positive cough stress test
* urgency score < stress score
* Patient's age between 40 - 65 years
* Desire to surgical correction of stress urinary incontinence or inadequate response to conservative treatment of SUI

Exclusion Criteria:

* Post-void residual volume >100cc
* Detrusor overactivity on preoperative multichannel urodynamic testing
* History of previous synthetic, biologic or fascial sub-urethral sling or any other surgery on external genitalia, bladder neck, bladder or urethra
* Desires future childbearing
* Chronic inguinal or vulvar abscess or history of Hidradenitis Suppurative
* History of bleeding diathesis or current anti-coagulation therapy
* Inguinal lymphadenopathy or inguinal/vulvar mass
* Current genitourinary fistula or urethral diverticulum
* Current sever cystocele or rectocele
* Active urinary infection
* Non-treated urge incontinency or any significant voiding dysfunction
* Neuromuscular disorders
* Uncontrolled Diabetes
* Reversible cause of incontinence (i.e. drug effect)
* Contraindications for surgery

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
24hr voiding diary reduction | 1 month
  Evaluation the 24hr voiding diary reduction by patient questionnaire 2hr pad test and cystourethroscopy and urodynamic.

SECONDARY OUTCOMES:
incontinence quality of life (I-Qol) | 1month
  Evaluation the increasing of incontinence quality of life (I-Qol) by questionnaire form.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine & Cell therapy center of Royan Institute; Farzaneh Sharifiaghdas, MD, Study Director — Urology and Nephrology Research Center, Shahid Beheshti University of Medical Sciences; Farshad Zohrabi, MD, Principal Investigator — Urology and Nephrology Research Center, Shahid Beheshti University of Medical Sciences; Reza Moghadasali, PhD, Principal Investigator — Department of Regenerative Medicine And Royan Cell Therapy Center Royan Institute For stem Cell Biology and Technology
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org